CLINICAL TRIAL: NCT03783884
Title: A Randomized, Controlled, Open-labeled, Multi-center Clinical Trial to Evaluate the Safe and Effective Performance of the Lungpacer Diaphragm Pacing Therapy System in Patients Who Have Failed to Wean From Mechanical Ventilation.
Brief Title: A Protocol Comparing Temporary Transvenous Diaphragm Pacing to Standard of Care for Weaning From Mechanical Ventilation
Acronym: RESCUE 3
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment rate.
Sponsor: Lungpacer Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P-300
Record Dates: First submitted 2018-12-19; First posted 2018-12-21 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Ventilator Induced Diaphragm Dysfunction
Keywords: VIDD; Diaphragm Atrophy; Weaning Failure; VLT; SBT; VILI; Phrenic Nerve Stimulation; Maximal Inspiratory Pressure

STUDY DESIGN:
Intervention Model Description: 1:1 randomization of treatment and control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Treatment (Active Comparator): Subject receives Lungpacer Catheter for transvenous phrenic nerve stimulation to deliver Diaphragm Pacing Therapy Sessions. DPT sessions are 6 sets of 10, delivered twice daily, for a total of 120 stimulation reps per day, plus standard of care for weaning from mechanical ventilation.
  Interventions: Device: Lungpacer Diaphragm Pacing Therapy
- Control (No Intervention): Subject does not receive Lungpacer Catheter or DPT. Subject receives only Standard of care for weaning from mechanical ventilation.

INTERVENTIONS:
Device: Lungpacer Diaphragm Pacing Therapy — Transvenous phrenic nerve stimulation to induce diaphragm contraction.
  Other Names: Lungpacer DPTS; AeroPace System
  Arms: Treatment

SUMMARY:
This clinical investigation is an open-label, multi-center RCT to demonstrate the safety and effective performance of the Lungpacer DPTS (plus standard of care) as compared to Control (standard of care only) in patients aged 18 years or older who are receiving mechanical ventilation. Eligible Subjects will have received mechanical ventilation for ≥96 hours (4 days) and have failed two weaning attempts.

The goal or outcome is to show a numerically greater proportion of subjects weaned in the Treatment (Lungpacer DPTS) group as compared to the Control group.

DETAILED DESCRIPTION:
The intended patient population is applicable for Lungpacer DPT because there are no noninvasive alternative treatments for patients who are difficult to wean from MV (i.e., ≥96 hours (4 days) on MV) or who have required prolonged MV (>7 days). The intended patient population includes approximately one-third of all patients on mechanical ventilation. Under standard of care, approximately 50% of these patients will recover from mechanical ventilation (Jung, 2016). Standard of care involves daily weaning attempts, known as Spontaneous Breathing Trials (SBTs) or Ventilator Liberation Trials (VLTs) that are intended to encourage diaphragm use and strengthening over time.Therefore, Lungpacer DPT efficacy evaluation must be compared to standard of care in a Control group. Lack of recovery from mechanical ventilation may be due to the inability of a patient to participate in VLTs or weaning attempts, due to extensive diaphragm weakness or sedation, the inability of VLTs to induce sufficient diaphragm strengthening, or co-morbidities that prevent recovery.

ELIGIBILITY:
Inclusion Criteria:

1. Are 18 years or older, and,
2. Have been mechanically ventilated for ≥96 hours (4 days), and,
3. Have satisfied the Readiness-to-Wean criteria, and,
4. Have failed at least 2 weaning attempts (that were conducted at least 48 hours after initiation of MV, and, that were conducted on different calendar days, and, at least one of which was the protocol-specific Ventilator Liberation Trial).

Exclusion Criteria:

1. MIP (absolute value) >50 cm H2O;
2. Invasive mechanical ventilation >90 days;
3. Currently on ECMO;
4. Weaning failure due to hypervolemia;
5. Medical history (including imaging) or known anatomy that prevents percutaneous insertion of the Catheter into the intended thoracic vein on the left side.
6. Clinically overt congestive heart failure that is preventing weaning;
7. Currently being treated with neuromuscular blockade;
8. Pre-existing neurological, neuromuscular or muscular disorder that could affect the respiratory muscles;
9. Pre-existing severe chronic pulmonary fibrosis;
10. Pleural effusions occupying greater than one third of the pleural space on either side;
11. BMI >45 kg/m2;
12. Known or suspected phrenic nerve paralysis;
13. Any electrical device (implanted or external) that may be prone to interaction with, or interference from the Lungpacer DPTS including neurological pacing/stimulator devices, cardiac pacemakers and defibrillators;
14. Current hemodynamic instability, sepsis or septic shock;
15. Prior bacteremia reported within the last 48 hours;
16. Anticipating withdrawal of life support and/or shift to palliation as the goal of care;
17. Known or suspected to be pregnant or lactating;
18. Currently being treated in another clinical trial studying an experimental treatment that could affect the study primary outcome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2019-06-14 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2023-01-27 (Actual)

PRIMARY OUTCOMES:
Successful Weaning | 30 days
  The proportion of subjects who are successfully weaned will be statistically significantly greater for subjects randomized to Treatment (Lungpacer DPTS) compared to subjects randomized to Control.
Adverse Event Profile | 30 days
  Characterize the adverse event profile to support an observed consistent risk profile for subjects randomized to Treatment compared to subjects randomized to Control.

SECONDARY OUTCOMES:
Days on MV | Successful weaning or Day 30
  The average days on mechanical ventilation from Day 1 to removal from MV associated with successful weaning or Day 30, whichever comes first, will be statistically significantly smaller for subjects randomized to Treatment as compared to subjects randomized to Control.
Maximal Inspiratory Pressure (MIP) Change | 30 days
  The mean improvement in inspiratory muscle strength as shown by the change in Maximal Inspiratory Pressure (MIP) from randomization to last available measure in subjects randomized to Treatment is superior to that in subjects randomized to Control.
Rapid Shallow Breathing Index (RSBI) Change | 30 days
  To determine change in Rapid Shallow Breathing Index (RSBI) from randomization to last available measure in subjects randomized to Treatment as compared to Control.
Mortality | 30 days
  To compare Treatment (Lungpacer DPTS) subjects to Control subjects for mortality through Day 30.

OTHER OUTCOMES:
Time to first successful Ventilator Liberation Trial (VLT) after randomization | Successful VLT or 30 days
  Assessment of time to first successful VLT in the Treatment group as compared to the Control group.
Cessations and re-instatements of MV through Day 30 or study exit. | 30 days
  Assessment of cessations and re-instatements of MV (e.g., reintubation) through Day 30 in the Treatment group as compared to the Control group.
Tracheotomy after randomization | 30 days
  Assessment of proportion of subjects tracheotomized from randomization (baseline) to Day 30 in the Treatment group as compared to the Control group.
Change in ventilator settings | 30 days
  Assessment of ventilator settings from baseline to last available measure in the Treatment group as compared to the Control group.
ICU admissions and discharges to Day 30. | 30 days
  Assessment of ICU admissions and discharges to Day 30 in the Treatment group as compared to the Control group.
Hospital admissions and discharges to Day 30. | 30 days
  Assessment of hospital admissions and discharges to Day 30 in the Treatment group as compared to the Control group.

CONTACTS AND LOCATIONS:
Locations (33):
- United States (22):
  - Stanford University Medical Center, Stanford, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - University of Florida, Shands, Gainesville, Florida
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - U of Illinois at Chicago, Chicago, Illinois
  - Edward Hines VA Hospital, Hines, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Indiana University Health Methodist Hospital, Indianapolis, Indiana
  - University of Louisville, Louisville, Kentucky
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - CHI Health Creighton University Medical Center - Bergan Mercy, Omaha, Nebraska
  - Englewood Hospital Medical Center, Englewood, New Jersey
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Kent County Memorial Hospital, Warwick, Rhode Island
  - Prisma Health Baptist Hospital, Columbia, South Carolina
  - University of Texas Southwestern, Zale Lipshy Hospital, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
- France (4):
  - CHU Angers, Angers
  - CHU Montpellier, Montpellier
  - Hôpital La Pitié-Salpêtrière, Paris
  - CHU Strasbourg, Strasbourg
- Germany (7):
  - Universitätsmedizin Greifswald, Greifswald, Mecklenburg-Vorpommern
  - Berlin Charite Mitte, Berlin
  - KEM Essen, Essen
  - SLK Löwenstein, Löwenstein
  - Nürnberg Klinikum Nord, Nuremberg
  - FKKG Schmallenberg, Schmallenberg
  - Solingen Krankenhaus Bethanien, Solingen

IPD SHARING:
Plan to Share IPD: No
Only investigators participating in this clinical trial will be able to see final de-identified participant data at the completion of the study.

REFERENCES:
- [Derived] Dres M, Ewert R, Conrad SA, Ataya A, Shrager J, Mortaza S, Delamaire F, Nilius G, Heine A, Mehta N, Ways J, Evans D, Paulon G, Khandwala F, Berry N, Viele K, Nelson T, Gilbertson M, Similowski T, Gama de Abreu M, Goligher EC; RESCUE-3 Trial Investigators. Temporary Transvenous Diaphragm Neurostimulation for Weaning from Mechanical Ventilation (RESCUE-3). Am J Respir Crit Care Med. 2025 Jun 11. doi: 10.1164/rccm.202505-1056OC. Online ahead of print. PMID 40498082
- See also: Sponsor website — http://lungpacer.com